CLINICAL TRIAL: NCT06465511
Title: Survivorship Intervention for Patients Living With Advanced and Metastatic Cancers: a Randomized Controlled Feasibility Study
Brief Title: Supportive Clinic for Patients Living With Advanced and Metastatic Cancers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW24-177
Record Dates: First submitted 2024-06-11; First posted 2024-06-20 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Physical Symptom Distress
Keywords: Physical symptom distress; self-efficacy in managing cancer; health-related quality of life; survivorship intervention; advanced cancer; randomised controlled trial; psychooncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a 2-arm feasibility trial study with an intervention group and a control group. Computer-generated block randomization sequences will be generated by a statistician who is blinded to the identity of participants prior to the start of the trial. A block randomisation structure with randomly permuted block sizes of 2 and 4 will be used to reduce selection bias and ensure close balance of the numbers in each arm. The serially labelled opaque sealed envelope method will be used for randomisation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to the intervention or the control arm.
  The participants are masked in terms of not knowing that the intervention are hypothesized to yield larger effects than the others (i.e. controls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive clinic (Experimental): Patients randomized to the intervention arm will attend a 120-minute survivorship clinic in which each participant will be assessed by members of a multidisciplinary team comprising an oncology nurse practitioner, a dietitian, a cancer exercise specialist, and a counsellor.
  Interventions: Behavioral: Supportive clinic
- Control: Self-management (Active Comparator): Patients randomized to the control group will be given a set of pamphlets explaining symptoms and describing skill-based self-management for symptom management and lifestyle recommendations.
  Interventions: Behavioral: Control: Self-management

INTERVENTIONS:
Behavioral: Supportive clinic — During the visit, each patient will receive a personalized feedback summary, including an assessment and recommendation on managing physical and psychological symptoms, an evaluation and recommendation on dietary advice, an assessment and recommendation on physical activity, and advice on managing potential psychosocial issues by the multidisciplinary team.
  Arms: Supportive clinic
Behavioral: Control: Self-management — Each pamphlet given to the patients addresses one of the 7 most commonly-reported symptoms (sleep difficulties, fatigue, neuropathy, pain, anxiety, depression, and fear of cancer progression) observed in Hong Kong patients with advanced or metastatic cancer, plus two on lifestyle recommendations (physical activity and eating well). All pamphlets are developed based on the self-management framework.
  Arms: Control: Self-management

SUMMARY:
To conduct a feasibility trial to examine the feasibility and acceptability of conducting a randomized controlled trial that evaluates the effect of the survivorship care intervention on patient-reported outcomes, defined as symptom distress and health-related quality of life.

DETAILED DESCRIPTION:
The primary aim of this study is to examine the feasibility and acceptability of conducting a randomized controlled trial (RCT) that evaluates a community-based survivorship care intervention to reduce symptom distress and improve health-related quality of life and self-management efficacy among patients with advanced or metastatic cancer. No hypothesis was proposed for this feasibility trial as the current Consolidation Standards of Reporting Trials (CONSORT) guidelines for reporting feasibility trials do not recommend hypothesis testing of clinical outcomes. The rationale is that pilot trials are often underpowered to detect differences, and this should be the aim of the main trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced or metastatic cancer
* are at least 18 years of age
* physically able to attend the supportive clinic.

Exclusion Criteria:

* Participants will be excluded from the study if they are non-Cantonese-, non-Mandarin-, or non-English-speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of subject recruitment | baseline
  number of participants consent and being randomized/number of eligible patients x 100
Rate of subject retention | baseline, 6-months and 9- months post-baseline
  number of participants who complete follow-up assessments at 6 and 9 months post-baseline/number of participants enrolled x 100
Adherence rate to intervention | immediate post-intervention
  number of participants who complete the intervention/number of being allocated to attend the intervention x 100
Rate of missing data | baseline, 6-months and 9- months post-baseline
  number of participants with completed datasets for outcome measures/number of participant enrolled x 100
Change of symptom distress | baseline, 6-months and 9- months post-baseline
  The 10-items Edmonton Symptom Checklist (ESAS) will be used to assess symptom distress. The ESAS assesses 10 symptoms commonly observed in cancer patients: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath, and sleep. A numerical rating scale 0 (no symptom at all) to 10 (the worst possible symptom) is used to measure distress associated with each symptom. ESAS has been widely adopted worldwide for standardized symptom screening in routine cancer care including palliative care, The total scores ranges from 0 to 100, with a higher score indicating greater total symptom distress. The minimal clinically important difference for improvement of the ESAS total symptom scores is 5.7 .
change of health-related quality of life | baseline, 6-months and 9- months post-baseline
  The Standard Chinese version of the European Organization Research Treatment Cancer (EORTC) general quality of life questionnaire (QLQ-C30) will assess health-related quality of life. The EORTC QLQ-C30 includes 30 items that measure five function scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health QoL subscale, five single symptom items (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and financial difficulty. All of the scales range in score from 0 to 100.The 10-point EORTC-QLQ-C30 scores changes are considered to be clinically important.

SECONDARY OUTCOMES:
Change of self-efficacy | baseline, 6-months and 9- months post-baseline
  Self-efficacy assessed by Self-Efficacy for Managing Chronic Disease scale (SEMCDS). This is a 6-item scale assessing patients' confidence to perform six self-management behaviours. Each item is rated on a 10-point Likert scale, with a total score ranging from 6 to 60. A high score indicates high self-efficacy. It has been used with cancer patients.
Change of supportive care needs | baseline, 6-months and 9- months post-baseline
  The Chines version of the 44-item Supportive Care Needs Survey for Partners and Caregivers (SCNS-P&C) will be used to assess caregiver support care needs. The SCNS-P&C assesses four domains of needs: Health care service needs, psychological and emotional needs, work and social needs, and information needs. Each item is rated on a 4-item scale (1= no need, 2 = low need, 3 = moderate need, and 4 = high need). A high score indicates greater unmet supportive care needs.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lam, Phd, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (5):
- Hong Kong (5):
  - Center of Cancer Medicine, Queen Mary Hospital, Hong Kong
  - JCICC, Hong Kong
  - Queen Mary Hospital-Department of Obstetrics & Gynaecology, Hong Kong
  - Queen Mary Hospital-Department of Oncology, Hong Kong
  - Queen Mary Hospital-Department of Surgery, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.